CLINICAL TRIAL: NCT05504278
Title: An Open-label, Multi-center Phase Ib/III Study Evaluating the Efficacy and Safety of IBI351 in Combination With Chemotherapy in Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Subjects With KRAS G12C Mutation
Brief Title: Efficacy and Safety of IBI351 in Combination With Chemotherapy in Advanced Non-squamous Non-small Cell Lung Cancer Subjects With KRAS G12C Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI351A301
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cetuximab; Pemetrexed; Carboplatin; sintilimab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IBI351 in combination with pemetrexed and cis-platinum/carboplatin (the subject with PD-L1 TPS<1%) (Experimental)
  Interventions: Drug: IBI351; Drug: pemetrexed; Drug: Carboplatin; Drug: cis-platinum
- IBI351 in combination with Cetuximab (Experimental)
  Interventions: Drug: IBI351; Drug: Cetuximab
- IBI351 monotherapy (Experimental)
  Interventions: Drug: IBI351
- IBI351 in combination with Sintilimab (Experimental)
  Interventions: Drug: IBI351; Drug: Sintilimab
- IBI351 in combination with pemetrexed and cis-platinum/carboplatin(the subject with PD-L1 TPS 1-49%) (Experimental)
  Interventions: Drug: IBI351; Drug: pemetrexed; Drug: Carboplatin; Drug: cis-platinum

INTERVENTIONS:
Drug: IBI351 — recommended dose, po
  Other Names: GFH925
Drug: Cetuximab — 500mg/m^2, Q2W, day1, i.v.
  Arms: IBI351 in combination with Cetuximab
Drug: pemetrexed — 500mg/m^2, Q3W, day1, i.v.
  Arms: IBI351 in combination with pemetrexed and cis-platinum/carboplatin (the subject with PD-L1 TPS<1%); IBI351 in combination with pemetrexed and cis-platinum/carboplatin(the subject with PD-L1 TPS 1-49%)
Drug: Carboplatin — AUC=5, Q3W, day1, i.v.
  Arms: IBI351 in combination with pemetrexed and cis-platinum/carboplatin (the subject with PD-L1 TPS<1%); IBI351 in combination with pemetrexed and cis-platinum/carboplatin(the subject with PD-L1 TPS 1-49%)
Drug: Sintilimab — 200mg, Q3W, day1, i.v.
  Other Names: IBI308
  Arms: IBI351 in combination with Sintilimab
Drug: cis-platinum — 75mg/m^2, Q3W, day1, i.v.
  Arms: IBI351 in combination with pemetrexed and cis-platinum/carboplatin (the subject with PD-L1 TPS<1%); IBI351 in combination with pemetrexed and cis-platinum/carboplatin(the subject with PD-L1 TPS 1-49%)

SUMMARY:
This Phase Ib/III study evaluates the efficacy and safety of IBI351 in combination with chemotherapy in advanced non-squamous NSCLC with KRAS G12C mutation.

DETAILED DESCRIPTION:
This Phase Ib/III study evaluates the efficacy and safety of IBI351 in combination with chemotherapy. There will be five cohorts of subjects, all of whom have KRAS G12C mutation and have advanced or metastatic NSCLC. Those five cohorts (A, B,C ,D and E) are treated with IBI351, IBI351+Sintilimab,IBI351+pemetrexed+cis-platinum/carboplatin,IBI351+Cetuximab, or IBI351+pemetrexed+cis-platinum/carboplatin respectively.

IBI351 is an orally available small molecule inhibitor of KRAS G12C.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of nonsquamous NSCLC with KRAS G12C mutation
2. Unresectable or metastatic disease
3. Adequate organ function
4. Not received any systemic antitumor therapy for locally advanced or metastatic non-squamous NSCLC previously.

Exclusion Criteria:

1. History of intestinal disease or major gastric surgery or inability to swallow oral medications
2. Prior therapy with agents targeting KRAS G12C mutation (e.g., AMG 510).
3. Active brain metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity | 12 months
  Number of participants with dose limiting toxicity in the dose escalation period
Evaluate clinical efficacy of IBI351 in combination with other therapeutic agents | 24 months
  Objective response rate per RECIST v1.1
Safety indicators during the introduction phase for IBI351 combination treatment : | 24 months
  Number of participants with Adverse events (AE), Treatment Emergent Adverse events (TEAE), treatment-related Adverse events (TEAE), TRAE) and the incidence of Serious Adverse events (SAE) (CTCAE v5.0 standard), with abnormal vital signs, abnormal physical exams, abnormal laboratory results and abnormal 12-lead electrocardiogram

SECONDARY OUTCOMES:
Evaluate plasma peak concentration of IBI351 | 12 months
  Cmax
Evaluate area under the plasma concentration-time curve (AUC) of IBI351 | 12 months
  AUC
Evaluate terminal half-life (t1/2) of IBI351 | 12 months
  t1/2
Evaluate clearance of IBI351 from the plasma | 12 months
  CL/F
Evaluate distribution of IBI351 | 12 months
  V/F
Evaluate clinical efficacy of IBI351 in combination with other therapeutic agents with other index | 24 months
  PFS, DCR,DOR, TTR per RECIST v1.1; OS
Number of subjects with adverse events of interest | 24 months
  AE
Number of subjects with treatment-related adverse events | 24 months
  TRAE
Number of subjects with serious adverse events | 24 months
  SAE
Number of subjects with treatment-emergent adverse events | 24 months
  TEAE
Overall Survival | 24 months
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Province Cancer Hospital, Jilin, Changchun, China